CLINICAL TRIAL: NCT01934790
Title: A Re-treatment Safety Study of Radium-223 Dichloride in Subjects With Castration-resistant Prostate Cancer With Bone Metastases Who Received an Initial Course of Six Doses of Radium-223 Dichloride 50 kBq/kg Every Four Weeks
Brief Title: Re-treatment Safety of Radium-223 Dichloride in Castration-resistant Prostate Cancer With Bone Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16506; 2013-003046-17 (EudraCT Number)
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Results first posted 2016-09-29 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radium-223 dichloride (Xofigo, BAY88-8223) (Experimental): Participants received intravenous (IV) injection of radium-223 dichloride 50 kBq/kg body weight every 4 weeks up to 6 injections.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Participants received intravenous (IV) injection of radium-223 dichloride 50 kBq/kg body weight every 4 weeks up to 6 injections.

SUMMARY:
Eligible subjects must have completed 6 doses of treatment of radium-223 dichloride and experienced no radium-223 dichloride-related SAEs (serious adverse events) or CTCAE (Common Terminology Criteria for Adverse Events) Grade 3 or 4 adverse event during or after the initial course of radium-223 dichloride that led to the discontinuation of treatment. 40 Subjects will be enrolled and will receive up to 6 doses of radium-223 dichloride 50 kBq/kg IV every 4 weeks.

The subject will be evaluated for AEs (adverse events) and laboratory tests at each visit every 4 weeks, prior to receiving radium-223 dichloride.

After the end of treatment visit the subjects will enter the active follow up period. Related AEs and SAEs and Lab tests will be evaluated at each visit every 4 weeks for the first 12 weeks, then every 12 weeks for up to 2 years after the last dose of radium-223 dichloride.

After the 2 years of active follow-up, subjects will enter the long-term follow-up period and will be followed via telephone follow-up at 6-month intervals for late toxicities and survival up to 7 years after the last dose of radium-223 dichloride or until death.

Joint safety reviews will regularly take place to oversee safety of the subjects conducted at regular intervals.

An interim analysis of the safety data will be conducted during the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate at any given point in time during disease history
* CRPC (castration-resistant prostate cancer) with clinical or radiologically confirmed bone progression
* Treatment with 6 injections of radium-223 dichloride 50 kBq/kg and no evidence of progression to bone (according to Prostate Cancer Clinical Trials Working Group 2 [PCWG2] criteria) during the first course of treatment
* Signed written informed consent prior to participating in any study related procedures. Willing and able to comply with the protocol, including follow-up visits and examinations

Exclusion Criteria:

* History of a radium-223 dichloride-related serious adverse event (SAE) or CTCAE Grade 3 or 4 adverse event (AE) during or after the initial course of radium-223 dichloride treatment that led to the discontinuation of treatment
* Less than 30 days from the last dose administered in the initial course of radium-223 dichloride treatment
* Visceral metastases 1 cm or greater in largest diameter and / or requiring local or systemic therapeutic intervention, as assessed by abdominal and pelvic magnetic resonance imaging (MRI) / computed tomography (CT) scan and / or chest X-ray within 30 days of the start of treatment
* Lymphadenopathy with lymph nodes exceeding 6 cm in short-axis diameter and / or requiring local or systemic therapeutic intervention. Enlarged lymph nodes of any size if the lymphadenopathy is thought to be a contributor to concurrent hydronephrosis.
* Current central nervous system (CNS) metastases
* Chronic conditions associated with non-malignant abnormal bone growth (e.g., confirmed Paget's disease of bone)
* Treatment with chemotherapy after the initial course of radium-223 dichloride treatment
* Prior hemibody external radiotherapy
* Prior systemic radiotherapy with strontium-89, samarium-153, rhenium-186, or rhenium-188
* Any other serious illness or medical conditions

  * Crohn's disease or ulcerative colitis
  * History of documented bone marrow dysplasia
  * Unmanageable fecal incontinence
* Imminent or established spinal cord compression based on clinical findings and / or MRI that has not yet been treated
* Other malignancy treated within the last 3 years (except non-melanoma skin cancer or low-grade superficial bladder cancer)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-12-22 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2017-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- United States (3):
  - New Orleans, Louisiana
  - Omaha, Nebraska
  - Syracuse, New York
- Kuopio, Finland
- Israel (4):
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
- Italy (2):
  - Forlì-Cesena, Emilia-Romagna
  - Milan, Lombardy
- Norway (2):
  - Bergen
  - Lørenskog
- Spain (3):
  - Córdoba, Andalusia
  - Barcelona
  - Málaga
- Umeå, Sweden

REFERENCES:
- [Derived] Sartor O, Heinrich D, Mariados N, Mendez Vidal MJ, Keizman D, Thellenberg Karlsson C, Peer A, Procopio G, Frank SJ, Pulkkanen K, Rosenbaum E, Severi S, Trigo J, Trandafir L, Wagner V, Li R, Nordquist LT. Re-treatment with radium-223: 2-year follow-up from an international, open-label, phase 1/2 study in patients with castration-resistant prostate cancer and bone metastases. Prostate. 2019 Oct;79(14):1683-1691. doi: 10.1002/pros.23893. Epub 2019 Aug 23. PMID 31442327
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 59 participants were screened in 7 countries worldwide, from 22-Dec-2013 (first patient first visit) to 12-Apr-2017 (last patient last visit).
Pre-assignment Details: The study was conducted at 16 study centers that screened 59 participants. Of them, 14 were screening failures and the remaining 45 participants were assigned to treatment.
Period: Treatment
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Started | 45 (Eligible for treatment)
Participants Received Study Treatment | 44
Completed | 29
Not Completed | 16
Not completed — Adverse Event | 3
Not completed — Clinical progression | 6
Not completed — Radiological progression | 4
Not completed — Withdrawal by Subject | 2
Not completed — Study drug never administered | 1
Period: Active Follow up
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Started | 34
Completed | 10
Not Completed | 24
Not completed — Death | 20
Not completed — Physician Decision | 2
Not completed — Progressive disease | 1
Not completed — Other reason | 1
Period: Long Term Follow up
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: Years] | 71 [52 to 91]
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 13
  >=65 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 44
Baseline Eastern Cooperative Oncology Group (ECOG) Performance status (PS) score [Number; unit: Participants] — Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is a scale that measures how cancer affects a patient. The scale ranges from 0 (fully active) to 5 (dead).
  Participants
    0 | 14
    1 | 27
    2 | 3
Number of bone lesions [Number; unit: Participants]
  1-5 | 18
  6-20 | 15
  > 20, not a superscan | 6
  Superscan | 5
Prostate specific antigen (PSA) - mean value [Mean (Standard Deviation); unit: microgram per liter] | 211.59 (452.84)
Total alkaline phosphatase (ALP) - mean value [Mean (Standard Deviation); unit: Unit per liter] | 122.60 (118.49)
Time from initial diagnosis of bone metastasis [Median (Full Range); unit: Months] | 43.12 [7.6 to 172.4]
Time from initial diagnosis [Median (Full Range); unit: Months] | 80.34 [11.8 to 287.9]
Time since initial treatment with radium-223 dichloride [Median (Full Range); unit: Months] | 6.05 [1.2 to 17.1]
Prostate specific antigen (PSA) - median value [Median (Full Range); unit: microgram per liter] | 67.66 [0.05 to 2349.04]
Total alkaline phosphatase (ALP) - median value [Median (Full Range); unit: Unit per liter] | 85 [29 to 705]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence (i.e., any unfavorable and unintended sign [including abnormal laboratory findings], symptom, or disease) in a participant or clinical investigation participant after providing written informed consent for participation in the study. A treatment-emergent adverse events (TEAE) is defined as any event arising or worsening after the start of study drug administration until 30 days after the last administration of radium-223 dichloride.
Time Frame: Up to 2.5 years
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Participants | 41

2. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: TESAE occurred after the start of radium-223 dichloride treatment until 30 days after the last dose and results in death; is life-threatening; requires inpatient hospitalization or prolongs existing hospitalization; results in persistent or significant disability or incapacity; is a congenital anomaly / birth defect; is another medically important serious event as judged by the investigator; or is an occurrence of leukemia, myelodysplastic syndrome, aplastic anemia, myelofibrosis, and primary bone cancer or any other new primary malignancy, such as acute myeloid leukemia.
Time Frame: Up to 2.5 years
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Participants | 13

3. Primary Outcome: Number of Participants With Radium-223 Dichloride-related AEs in the Active Follow-up Period
Description: An adverse event (AE) is any untoward medical occurrence (i.e., any unfavorable and unintended sign [including abnormal laboratory findings], symptom, or disease) in a participant or clinical investigation participant after providing written informed consent for participation in the study.
Time Frame: Up to 2 years after last treatment
Population: Active Follow-up Analysis Set: participants who were reported in the End of Treatment (EOT) electronic case report form (eCRF) as planning to participate in the active follow-up.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 34
Participants | 1

4. Primary Outcome: Number of Participants With Radium-223 Dichloride-related SAEs in the Active Follow-up Period
Description: Treatment-related SAE is any SAE that, according to the investigator's causality assessment, is possibly or probably related to treatment with radium-223 dichloride.
Time Frame: Up to 2 years after last treatment
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 34
Participants | 0

5. Primary Outcome: Number of Participants With High/Low Abnormalities in Hematology Variables at Any Visit After Treatment Start
Time Frame: Up to 2.5 years
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Participants
  Eosinophils (GIGA/L) - High | 1
  Ery. Mean Corpuscular HGB Conc. (g/dL) - High | 1
  Ery. Mean Corpuscular Hemoglobin (pg) - High | 16
  Ery. Mean Corpuscular Volume (fL) - High | 22
  Leukocytes (GIGA/L) - High | 5
  Monocytes (GIGA/L) - High | 7
  Neutrophils (GIGA/L) - High | 9
  Platelets (GIGA/L) - High | 1
  Basophils (GIGA/L) - Low | 2
  Eosinophils (GIGA/L) - Low | 7
  Ery. Mean Corpuscular HGB Conc. (g/dL) - Low | 17
  Ery. Mean Corpuscular Hemoglobin (pg) - Low | 4
  Ery. Mean Corpuscular Volume (fL) | 3
  Erythrocytes (T/L) - Low | 43
  Hematocrit (%) - Low | 43
  Hemoglobin (g/dL) - Low | 43
  Leukocytes (GIGA/L) - Low | 21
  Lymphocytes (GIGA/L) - Low | 36
  Monocytes (GIGA/L) - Low | 2
  Neutrophils (GIGA/L) - Low | 10
  Platelets (GIGA/L) - Low | 11

6. Primary Outcome: Number of Participants With High/Low Abnormalities in Biochemistry Variables at Any Visit After Treatment Start
Time Frame: Up to 2.5 years
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Participants
  Alanine Aminotransferase (U/L) - High | 2
  Alkaline Phosphatase (U/L) - High | 14
  Aspartate Aminotransferase (U/L) - High | 6
  Bilirubin (mg/dL) - High | 1
  Creatinine (mg/dL) - High | 7
  Sodium (mmol/L) - High | 6
  Alanine Aminotransferase (U/L) - Low | 4
  Albumin (g/dL) - Low | 10
  Aspartate Aminotransferase (U/L) - Low | 1
  Bilirubin (mg/dL) - Low | 4
  Creatinine (mg/dL) - Low | 7
  Sodium (mmol/L) - Low | 14

7. Primary Outcome: Number of Participants Who Discontinued Radium-223 Dichloride Treatment Due to Treatment Emergent AEs or Death
Description: as for outcome 1
Time Frame: Up to 2.5 years
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Participants | 2

8. Other Pre Specified Outcome: Radiological Progression Free Survival (rPFS)
Description: Radiological progression-free survival (rPFS) was defined as the time from the treatment start date to the date of radiological disease progression or death from any cause (if death occurred before such progression), as documented by the investigator. Participants not experiencing death or radiological disease progression at the database cutoff for primary completion were censored at the last radiological disease progression assessment.
Time Frame: Up to 2 years after last treatment
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Months | 9.9 [6.9 to 12.9]

9. Other Pre Specified Outcome: Time to Radiological Bone Progression
Description: Time to radiological bone progression was defined as the time (days) from the treatment start date to the date of radiological bone progression (according to the adapted PCWG2 [Prostate Cancer Clinical Trials Working Group 2] criteria), as documented by the investigator. Participants not experiencing radiological bone progression at the database cutoff for primary completion were censored at the last radiological bone progression assessment.
Time Frame: Up to 2 years after last treatment
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Months | NA [9.9 to NA] — value could not be estimated due to censored values

10. Other Pre Specified Outcome: Percentage of Participants With Total Alkaline Phosphatase (ALP) Response
Description: Total alkaline phosphatase (ALP) response was defined as ≥ 30% reduction of the blood total ALP level compared with the baseline values. Total ALP response rate was defined as the number of participants with total ALP response divided by the total number of participants evaluable for total ALP response.
Time Frame: Up to 2.5 years
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Percentage of participants
  12 Week: number analyzed (Participants) | 33
  12 Week | 39.4 [22.9 to 57.9]
  24 Week: number analyzed (Participants) | 36
  24 Week | 30.6 [16.3 to 48.1]
  Anytime | 43.2 [28.3 to 59.0]

11. Other Pre Specified Outcome: Time to Total ALP Progression
Description: Total ALP progression was defined as a ≥ 25% increase above the nadir (lowest baseline or post-baseline) value to at least 1.5 x ULN (upper limit of normal). The time to total ALP progression was defined as the time (days) from the treatment start date to the date of first total ALP progression. Participants not experiencing ALP progression at the database cutoff date, whether or not surviving, were censored at the last ALP laboratory assessment.
Time Frame: Up to 2 years after last treatment
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Months | NA [11.9 to NA] — value could not be estimated due to censored values

12. Other Pre Specified Outcome: Percent Change in Total ALP
Time Frame: Baseline and Week 12, Week 24
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Percent change
  Week 12: number analyzed (Participants) | 33
  Week 12 | -17.1 (32.74)
  Week 24: number analyzed (Participants) | 36
  Week 24 | -15.0 (35.10)

13. Other Pre Specified Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response
Description: Prostate specific antigen (PSA) response was defined as a ≥ 30% reduction of blood PSA level compared with the baseline value, confirmed by a second subsequent PSA value with a ≥ 30% reduction from baseline approximately 4 or more weeks later. Prostate specific antigen response rate was defined as the number of participants with PSA response divided by the total number of participants evaluable for PSA response.
Time Frame: Up to 2.5 years
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Percentage of participants
  12 Week: number analyzed (Participants) | 32
  12 Week | 6.3 [0.8 to 20.8]
  24 Week: number analyzed (Participants) | 36
  24 Week | 0 [0 to 9.7]
  Anytime | 9.1 [2.5 to 21.7]

14. Other Pre Specified Outcome: Time to PSA Progression
Description: Prostate specific antigen progression was defined as a ≥ 25% increase above the nadir (lowest baseline or post-baseline) value, and an increase in absolute value of ≥ 2 ng/mL above nadir. The time to PSA progression was defined as the time (days) from the treatment start date to the date of first PSA progression. Participants without PSA progression as of the database cutoff for primary completion, whether or not surviving, were censored at the last PSA laboratory assessment.
Time Frame: Up to 2 years after last treatment
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Months | 2.2 [1.8 to 3.1]

15. Other Pre Specified Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time (days) from the treatment start date to the date of death due to any cause. For participants who were still alive or who were lost to follow-up as of the database cutoff date for the primary completion, OS was censored at the last known alive date on or prior to the database cutoff date.
Time Frame: Up to 2 years after last treatment
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Months | 24.4 [14.9 to 28.6]

16. Other Pre Specified Outcome: Percentage of Participants With Pain Improvement
Description: Pain improvement was defined in evaluable participants (participants with worst pain score [WPS] of 4 at baseline) as a 30% and 2-point decrease in WPS over 2 consecutive measurements conducted at least 4 weeks apart, without an increase in pain management. Pain improvement rate was the number of participants with pain improvement, divided by the total number of evaluable participants WPS was the mean of the WPS in the last 24 hours from the preceding 7 days.
Time Frame: Up to 2.5 years
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Percentage of participants
  12 Week: number analyzed (Participants) | 6
  12 Week | 0 [0 to 45.9]
  24 Week: number analyzed (Participants) | 8
  24 Week | 0 [0 to 36.9]
  Anytime: number analyzed (Participants) | 12
  Anytime | 8.3 [0.2 to 38.5]

17. Other Pre Specified Outcome: Time to Pain Progression
Description: Pain progression was defined in participants evaluable for pain progression at baseline, i.e., participants with a WPS of ≤ 7 at the baseline assessment. Pain assessment occurred daily for 1 week, beginning 1 week prior to each visit and including the day of the visit. An evaluable pain assessment interval required completion of a minimum of 4 out of 7 daily questions. Pain progression was defined as the occurrence of either a pain increase or an increase in pain management with respect to baseline, whichever occurred first.
Time Frame: Up to 2.5 years
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Months | NA [NA to NA] — value could not be estimated due to censored values

18. Other Pre Specified Outcome: Time to First Symptomatic Skeletal Event (SSE)
Description: Time to first symptomatic skeletal event (SSE) is the time (days) from the treatment start date to the first SSE on or following the start date. Participants not experiencing an SSE at the database cutoff date for primary completion, whether or not surviving, were censored at the last assessment for SSEs.
Time Frame: Up to 2 years after last treatment
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Months | 16.7 [9.7 to NA] — value could not be estimated due to censored values

19. Other Pre Specified Outcome: SSE-free Survival
Description: The SSE-FS is the time (days) from the treatment start date to the first SSE on or following the start date or death, whichever occurred first. Participants not experiencing death or an SSE at the database cutoff date for primary completion were censored at the last assessment for SSEs.
Time Frame: Up to 2 years after last treatment
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Months | 12.8 [9.5 to 24.4]

20. Post Hoc Outcome: Number of Participants With New SSE Related AEs During the Follow-up Period
Time Frame: Up to 2 years after last treatment
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 34
Participants | 0

21. Post Hoc Outcome: Number of Participants With New Primary Malignancies During Study Treatment or Follow-up Period
Time Frame: Up to 2 years after last treatment
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 34
Participants | 1

22. Post Hoc Outcome: Number of Deaths During Study Treatment or Follow-up Period
Time Frame: Up to 2 years after last treatment
Population: Safety Analysis Set (SAF): all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 44
Participants
  During Treatment Period | 1
  During Active follow-up Period | 23
  During Long-term follow-up Period | 4

23. Post Hoc Outcome: Number of Participants With Significant Meaningful Changes for Clinical Laboratory NCI-CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) Toxicity Grades During the Follow-up Period
Time Frame: Up to 2 years after last treatment
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 34
Participants | 0

24. Post Hoc Outcome: Number of Participants With Body Weight Changes During the Follow-up Period
Description: Participants were counted once during active follow-up for both increases (using the maximum body weight) and decreases (using the minimum body weight).
Time Frame: Up to 2 years after last treatment
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 34
Participants
  Increases < 5% | 23
  Increases 5-10% | 4
  Increases > 10% | 0
  Decreases < 5% | 13
  Decreases 5-10% | 9
  Decreases > 10% | 5

25. Post Hoc Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Score Worsened to >=3 During the Follow-up Period
Time Frame: Up to 2 years after last treatment
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Number analyzed (Participants) | 34
Participants | 4

ADVERSE EVENTS:
Time Frame: From start of study treatment until 30 days after last dose of study medication up to 2.5 years
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223)
Serious Adverse Events (participants affected / at risk) | 13/44
Other Adverse Events (participants affected / at risk) | 35/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 Dichloride (Xofigo, BAY88-8223) (N=44)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 2 (2)
Stomatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 Dichloride (Xofigo, BAY88-8223) (N=44)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 9 (11)
Nausea (Gastrointestinal disorders) | 11 (13)
Vomiting (Gastrointestinal disorders) | 5 (8)
Asthenia (General disorders) | 4 (4)
Fatigue (General disorders) | 12 (12)
Oedema peripheral (General disorders) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 5 (8)
White blood cell count decreased (Investigations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 8 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
Hypertension (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12-18 months after database lock at the earliest. Bayer will have 30-45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable). No publication of single center data should be done prior of publication if multi-center data.